CLINICAL TRIAL: NCT00953758
Title: A PHASE 1 STUDY TO EVALUATE THE SAFETY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF PF-04449913, AN ORAL HEDGEHOG INHIBITOR, ADMINISTERED AS SINGLE AGENT IN SELECT HEMATOLOGIC MALIGNANCIES
Brief Title: A Study Of PF-04449913 In Select Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B1371001; 2009-011285-29 (EudraCT Number)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-11

CONDITIONS: Hematologic Malignancies
Keywords: Chronic Myeloid Leukemia Myelofibrosis Myelodysplastic Syndrome Acute myeloid Leukemia Hedgehog inhibitor
MeSH Terms: conditions — Hematologic Neoplasms | interventions — glasdegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-04449913

INTERVENTIONS:
Drug: PF-04449913 — Escalating doses of PF-04449913 administered as tablets PO QD continuously in 28 day cycles

SUMMARY:
This study examines the effect of a small molecule inhibitor to the Sonic Hedgehog pathway on select hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with select advanced hematologic malignancies who are refractory, resistant or intolerant to prior therapies. They may be newly diagnosed and previously untreated, but not eligible for standard treatment options, or for whom standard therapies are not anticipated to result in a durable response.
* ECOG performance status 0 to 2
* Adequate organ function

Exclusion Criteria:

* Patients with active CNS disease
* Patient with active malignancy with the exception of basal cell carcinoma, non melanoma skin cancer, carcinoma in situ cervical or skin cancer
* Active GVHD other than Grade 1 skin involvement
* Known malabsorption syndrome
* Patient has an active, life threatening or clinically significant uncontrolled systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-03-03 (Actual); Primary Completion 2012-09-26 (Actual); Study Completion 2013-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (5):
  - UCSD Medical Center - La Jolla, La Jolla, California
  - Moores UCSD Cancer Center, La Jolla, California
  - UCSD Medical Center - Hillcrest, San Diego, California
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle Cancer Care Alliance, Seattle, Washington
- U.O. di Ematologia, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Fostvedt LK, Shaik N, Martinelli G, Wagner AJ, Ruiz-Garcia A. Exposure-response modeling of the effect of glasdegib on cardiac repolarization in patients with cancer. Expert Rev Clin Pharmacol. 2021 Jul;14(7):927-935. doi: 10.1080/17512433.2021.1925538. Epub 2021 May 18. PMID 33993815
- [Derived] Martinelli G, Oehler VG, Papayannidis C, Courtney R, Shaik MN, Zhang X, O'Connell A, McLachlan KR, Zheng X, Radich J, Baccarani M, Kantarjian HM, Levin WJ, Cortes JE, Jamieson C. Treatment with PF-04449913, an oral smoothened antagonist, in patients with myeloid malignancies: a phase 1 safety and pharmacokinetics study. Lancet Haematol. 2015 Aug;2(8):e339-46. doi: 10.1016/S2352-3026(15)00096-4. Epub 2015 Jul 26. PMID 26688487
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1371001&StudyName=A%20Study%20Of%20PF-04449913%20In%20Select%20Hematologic%20Malignancies

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04449913 5 mg: Participants received oral single agent PF-04449913 tablets 5 milligram (mg) once on Day -6 (as a lead-in dose), followed by once daily (QD) dosing starting from Cycle 1 Day 1, without interruption, in 28-day cycles (maximum duration: 537 days).
- PF-04449913 10 mg: Participants received oral single agent PF-04449913 tablets 10 mg once on Day -6 (as a lead-in dose), followed by QD dosing from Cycle 1 Day 1, without interruption, in 28-day cycles (maximum duration: 537 days).
- PF-04449913 20 mg: Participants received oral single agent PF-04449913 tablets 20 mg once on Day -6 (as a lead-in dose), followed by QD dosing starting from Cycle 1 Day 1, without interruption, in 28-day cycles (maximum duration: 537 days).
- PF-04449913 40 mg: Participants received oral single agent PF-04449913 tablets 40 mg once on Day -6 (as a lead-in dose), followed by QD dosing starting from Cycle 1 Day 1, without interruption, in 28-day cycles (maximum duration: 537 days).
- PF-04449913 80 mg: Participants received oral single agent PF-04449913 tablets 80 mg once on Day -6 (as a lead-in dose), followed by QD dosing starting from Cycle 1 Day 1, without interruption, in 28-day cycles (maximum duration: 537 days).
- PF-04449913 120 mg: Participants received oral single agent PF-04449913 tablets 120 mg once on Day -6 (as a lead-in dose), followed by QD dosing starting from Cycle 1 Day 1, without interruption, in 28-day cycles (maximum duration: 537 days).
- PF-04449913 180 mg: Participants received oral single agent PF-04449913 tablets 180 mg once on Day -6 (as a lead-in dose), followed by QD dosing starting from Cycle 1 Day 1, without interruption, in 28-day cycles (maximum duration: 537 days).
- PF-04449913 270 mg: Participants received oral single agent PF-04449913 tablets 270 mg once on Day -6 (as a lead-in dose), followed by QD dosing starting from Cycle 1 Day 1, without interruption, in 28-day cycles (maximum duration: 537 days).
- PF-04449913 400 mg: Participants received oral single agent PF-04449913 tablets 400 mg once on Day -6 (as a lead-in dose), followed by QD dosing starting from Cycle 1 Day 1, without interruption, in 28-day cycles (maximum duration: 537 days).
- PF-04449913 600 mg: Participants received oral single agent PF-04449913 tablets 600 mg once on Day -6 (as a lead-in dose), followed by QD dosing starting from Cycle 1 Day 1, without interruption, in 28-day cycles (maximum duration: 537 days).
Period: Overall Study
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Started | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5
Completed | 1 | 3 | 2 | 2 | 2 | 2 | 2 | 1 | 6 | 4
Not Completed | 2 | 0 | 2 | 2 | 6 | 1 | 1 | 4 | 3 | 1
Not completed — Death | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 3 | 1 | 0
Not completed — Participant refused further follow-up | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant went for transplant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg | Total
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 1 | 2 | 2 | 1 | 2 | 5 | 0 | 15
  >=65 years | 2 | 3 | 3 | 3 | 6 | 1 | 2 | 3 | 4 | 5 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 2 | 3 | 1 | 0 | 2 | 2 | 3 | 19
  Male | 1 | 2 | 1 | 2 | 5 | 2 | 3 | 3 | 7 | 2 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Cycle Dose-limiting Toxicities (DLTs)
Description: Any DLT event in Cycle 1: 1) Grade >=3 non-hematologic toxicity that had been maximally treated, 2) prolonged myelosupression that lasted greater than (>) 42 days from the point of detection in a normal bone marrow (less than [<] 500 per microliter [/uL] or platelet count <10,000/uL, or hemoglobin <8 gram per deciliter [g/dL] with <5% blasts and no evidence of disease or dysplasia), 3) inability to deliver >= 80% of the planned doses due to PF-04449913 related non-hematologic and hematologic toxicities
Time Frame: Cycle 1 Day 1 to end of Cycle 1 (28 days)
Population: Only participants who did not have major treatment deviations in Cycle 1 were evaluable for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 6 | 3 | 3 | 3 | 7 | 5
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (AEs) by National Cancer Institute (NCI) Common Terminology Criteria (CTC) for AEs (CTCAE) (Version 3.0) Grade
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs are events which occurred between first dose of study drug and 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. If the same participant in a given treatment had more than 1 occurrence in the same preferred term event category, only the worst CTCAE grade (1 = mild AE, 2 = moderate AE, 3 = severe AE, 4 = life-threatening or disabling AE, 5 = death related to AE) was reported.
Time Frame: Baseline up to 28 days post last dose of study medication (maximum duration: 537 days)
Population: The safety analysis set consisted of all enrolled participants who received at least 1 dose of PF-04449913, including the lead-in dose.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5
percentage of participants
  Any AEs, Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Any AEs, Grade 2 | 0.0 | 0.0 | 0.0 | 25.0 | 12.5 | 33.3 | 33.3 | 40.0 | 0.0 | 40.0
  Any AEs, Grade 3 | 0.0 | 66.7 | 50.0 | 25.0 | 50.0 | 33.3 | 66.7 | 20.0 | 55.6 | 20.0
  Any AEs, Grade 4 | 66.7 | 33.3 | 25.0 | 25.0 | 25.0 | 0.0 | 0.0 | 0.0 | 22.2 | 40.0
  Any AEs, Grade 5 | 33.3 | 0.0 | 12.5 | 25.0 | 12.5 | 33.3 | 0.0 | 40.0 | 22.2 | 0.0

3. Secondary Outcome: Percentage of Participants With Treatment-related Adverse Events (AEs), by NCI CTCAE Version 3.0) Grade
Description: An AE was any untoward medical occurrence in a participant. Treatment-related AEs are events that were assessed by the investigator as related to study medication. If the same participant in a given treatment had more than 1 occurrence in the same preferred term event category, only the worst CTCAE grade (1 = mild AE, 2 = moderate AE, 3 = severe AE, 4 = life-threatening or disabling AE, 5 = death related to AE) was reported.
Time Frame: Baseline up to 28 days post last dose of study medication (maximum duration: 537 days)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5
percentage of participants
  Any AEs, Grade 1 | 0.0 | 0.0 | 25.0 | 25.0 | 12.5 | 33.3 | 33.3 | 0.0 | 11.1 | 0.0
  Any AEs, Grade 2 | 0.0 | 0.0 | 0.0 | 50.0 | 12.5 | 0.0 | 0.0 | 80.0 | 33.3 | 20.0
  Any AEs, Grade 3 | 0.0 | 66.7 | 0.0 | 25.0 | 0.0 | 0.0 | 0.0 | 0.0 | 33.3 | 40.0
  Any AEs, Grade 4 | 33.3 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0 | 0.0 | 0.0 | 0.0 | 20.0
  Any AEs, Grade 5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Number of Participants With Vital Signs Values Meeting Categorical Summarization Criteria
Description: Participants with systolic blood pressure (BP) less than (<) 90 millimeters of mercury (mmHg), maximum increase and decrease from baseline systolic BP of more than or equal to (>=) 30 mmHg, diastolic BP <50 mmHg, maximum increase and decrease from baseline diastolic BP >=20 mmHg, and a heart rate of more than (>) 120 beats per minute (bpm) at any time post dose were summarized.
Time Frame: Screening up to maximum of 537 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5
Participants
  Systolic BP <90 mmHg | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Decrease from baseline systolic BP >=30 mmHg | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 1 | 2 | 1
  Increase from baseline systolic BP >=30 mmHg | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 1
  Diastolic BP <50 mmHg | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Decrease from baseline diastolic BP >=20 mmHg | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 3 | 0
  Increase from baseline diastolic BP >=20 mmHg | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 1
  Heart rate >120 bpm at any time post dose | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0

5. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Number of participants with laboratory test abnormalities without regard to baseline abnormality as per the pre defined criteria were reported. Laboratory test parameters included hematology, coagulation, liver function, renal function, electrolytes, clinical chemistry, and urinalysis (dipstick and microscopy).
Time Frame: Screening to EOT (maximum duration: 537 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5
Participants | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5

6. Secondary Outcome: Hedgehog Biomarker Modulation: Relative GLI1 Gene Expression to Baseline for Normal Skin on Cycle 1 Day 21
Description: Ribonucleic acid (RNA) was extracted from skin samples and complementary deoxyribonucleic acid (cDNA) was prepared. Gene expression was measured using custom Taqman low density array (TLDA) cards run on the Applied Biosystems ViiATM 7 system.
Time Frame: Baseline, Cycle 1 Day 21
Population: The pharmacodynamic (PD) analysis population included all enrolled participants who received at least 1 dose of PF-04449913 and had at least 1 PD parameter in at least 1 treatment period. Results were not collected and reported for the other reporting arms since none of the participants in those arms had evaluable PD samples.
Measure: Number; unit: ratio
Arm/Group | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg
Number analyzed (Participants) | 1 | 1 | 1
ratio | 0.1 | 0.0 | 0.0

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) on Lead-in
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24, 48, 96 and 120 hours post-dose during the lead-in period (Day -6)
Population: The pharmacokinetic (PK) analysis set included all enrolled and treated (received at least 1 dose of study medication) participants who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5
nanogram/milliliter (ng/mL) | 32.9 (3.0) | 59.0 (21) | 247 (47) | 313 (51) | 746 (56) | 1418 (22) | 1409 (79) | 1534 (72) | 3714 (30) | 4527 (64)

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) on Cycle 1 Day 21
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle 1 Day 21
Population: PK analysis set included all enrolled and treated (received at least 1 dose of study medication) participants who had at least 1 of the PK parameters of interest. N = the number of participants analyzed for Cycle 1. 1 participant from the 270-mg arm had dose reduction to 180 mg and is analyzed and reported under the 180-mg arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 4 | 2 | 6 | 4
ng/mL | 45.4 (12) | 75.0 (30) | 249 (35) | 565 (83) | 871 (35) | 1621 (10) | 2069 (41) | 1504 (NA) — Geometric coefficient of variation (%CV) not reported when there are 2 or less participants. | 4989 (7.0) | 6413 (65)

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Lead-in
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24, 48, 96 and 120 hours post-dose during the lead-in period (Day -6)
Population: The PK analysis set included all enrolled and treated (received at least 1 dose of study medication) participants who had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5
hours | 2.0 [1.0 to 4.0] | 2.0 [1.2 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 4.0] | 2.0 [1.3 to 4.0] | 2.0 [1.1 to 4.0] | 2.0 [1.0 to 4.1] | 2.0 [1.3 to 4.5] | 2.0 [1.1 to 4.0]

10. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Cycle 1 Day 21
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle 1 Day 21
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 4 | 2 | 6 | 4
hours | 2.2 [1.0 to 4.0] | 1.0 [1.0 to 2.0] | 0.92 [0.92 to 1.0] | 1.0 [1.0 to 2.0] | 1.3 [1.0 to 2.0] | 2.2 [2.0 to 6.1] | 1.1 [1.0 to 2.0] | 3.1 [2.13 to 4.07] | 4.0 [1.1 to 4.2] | 3.2 [2.2 to 4.6]

11. Secondary Outcome: Apparent Oral Clearance (CL/F) on Lead-in
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24, 48, 96 and 120 hours post-dose during the lead-in period (Day -6)
Population: The PK analysis set included all enrolled and treated (received at least 1 dose of study medication) participants who had at least 1 of the PK parameters of interest. N = number of participants with available data for this PK parameter in this period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)/hour
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 7 | 3 | 3 | 5 | 8 | 5
liter (L)/hour | 7.61 (19) | 12.7 (23) | 5.63 (50) | 11.1 (37) | 9.13 (64) | 8.33 (36) | 8.48 (64) | 10.8 (110) | 5.90 (19) | 6.93 (58)

12. Secondary Outcome: Apparent Oral Clearance (CL/F) on Cycle 1 Day 21
Description: as for outcome 11
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle 1 Day 21
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 4 | 2 | 6 | 4
L/hour | 8.57 (9.0) | 13.3 (27) | 7.79 (13) | 6.52 (62) | 10.7 (46) | 5.33 (13) | 7.81 (48) | 11.8 (NA) — As planned, Geometric CV cannot be calculated and reported when the number of participants is 2 or less. | 5.68 (24) | 8.36 (51)

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F) on Lead-in
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24, 48, 96 and 120 hours post-dose during the lead-in period (Day -6)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 7 | 3 | 3 | 5 | 8 | 5
liter (L) | 262 (32) | 455 (41) | 265 (62) | 367 (38) | 292 (71) | 316 (52) | 210 (92) | 359 (143) | 185 (50) | 191 (78)

14. Secondary Outcome: Plasma Decay Half-life (t1/2) on Lead-in
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24, 48, 96 and 120 hours post-dose during the lead-in period (Day -6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 7 | 3 | 3 | 5 | 8 | 5
hours | 25.1 (9.6) | 25.1 (4.3) | 34.3 (14) | 23.3 (4.2) | 23.3 (8.1) | 26.5 (4.0) | 17.4 (3.3) | 23.6 (5.5) | 23.9 (14) | 19.6 (4.7)

15. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Infinity (AUCinf) on Lead-in
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24, 48, 96 and 120 hours post-dose during the lead-in period (Day -6)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 7 | 3 | 3 | 5 | 8 | 5
nanograms*hour/milliliter (ng*hr/mL) | 657 (19) | 786 (23) | 3548 (50) | 3614 (38) | 8755 (64) | 14430 (35) | 21280 (64) | 25110 (109) | 67720 (19) | 86620 (58)

16. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) on Cycle 1 Day 21
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle 1 Day 21
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 4 | 2 | 6 | 4
ng*hour/mL | 583 (10) | 753 (27) | 2566 (13) | 6134 (61) | 7482 (46) | 22520 (13) | 23060 (47) | 22990 (NA) — Not reported when the number of participants is 2 or less. | 70430 (24) | 71710 (51)

17. Secondary Outcome: Average Plasma Concentration (Cavg) on Cycle 1 Day 21
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle 1 Day 21
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 4 | 2 | 6 | 4
ng/mL | 24.3 (9.0) | 31.4 (27) | 107 (13) | 256 (61) | 312 (46) | 940 (13) | 961 (48) | 960 (NA) — Not reported when the number of participants is 2 or less. | 2933 (24) | 2986 (51)

18. Secondary Outcome: Minimum Plasma Concentration (Cmin) on Cycle 1 Day 21
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle 1 Day 21
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 4 | 2 | 6 | 4
ng/mL | 14.7 (15) | 18.9 (14) | 54.7 (46) | 162 (107) | 116 (48) | 360 (115) | 408 (42) | 428 (NA) — Not reported when the number of participants is 2 or less. | 1113 (44) | 1641 (59)

19. Secondary Outcome: Pre-dose Concentration (Ctrough) on Cycle 1 Day 21
Time Frame: Pre-dose on Cycle 1 Day 21
Population: PK analysis set included all enrolled and treated (received at least 1 dose of study medication) participants who had at least 1 of the PK parameters of interest. N = number of participants with available data for this parameter in this period. 1 participant from the 270-mg arm had dose reduction to 180 mg and is analyzed and reported under 180-mg.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 5 | 3 | 4 | 2 | 7 | 3
ng/mL | 15.1 (17) | 18.9 (14) | 67.8 (48) | 170 (121) | 120 (53) | 495 (56) | 485 (86) | 428 (NA) — Not reported when the number of participants is 2 or less. | 1291 (42) | 1871 (57)

20. Secondary Outcome: Accumulation Ratio (Rac)
Description: Accumulation ratio was calculated as AUCtau at steady state (Cycle 1/Day 21)/AUCtau on Cycle 1 Day 1.
Time Frame: Pre-dose, 1 hour post-dose on Cycle 1 Day 1; Pre-dose, 0.5, 1, 2, 4, 8 and 24 hours post-dose on Cycle 1 Day 21
Population: as for outcome 8
Measure: Median (Full Range); unit: ratio
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 4 | 2 | 6 | 4
ratio | 1.4 [1.3 to 1.7] | 1.6 [1.1 to 1.8] | 1.6 [1.6 to 1.9] | 2.4 [2.3 to 3.0] | 1.4 [1.1 to 2.2] | 2.5 [1.5 to 3.4] | 1.4 [0.8 to 2.0] | 1.5 [0.5 to 2.6] | 1.2 [1.0 to 2.8] | 1.4 [1.1 to 1.6]

21. Secondary Outcome: Linearity Ratio (Rss)
Description: Linearity ratio was calculated as AUCtau at steady state (Cycle 1/Day 21)/AUCinf after single dose (Lead-in Period [Day -6]).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24, 48, 96, 120 hours post-dose during the lead-in period (Day -6); Pre-dose, 0.5, 1, 2, 4, 8 and 24 hours post-dose on Cycle 1 Day 21
Population: as for outcome 8
Measure: Median (Full Range); unit: ratio
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 3 | 4 | 2 | 6 | 4
ratio | 0.91 [0.79 to 0.98] | 1.1 [0.70 to 1.2] | 0.76 [0.71 to 1.2] | 1.6 [1.5 to 2.2] | 0.97 [0.75 to 1.7] | 2.1 [0.91 to 2.1] | 1.0 [0.5 to 1.4] | 1.0 [0.30 to 1.77] | 0.86 [0.76 to 2.1] | 0.97 [0.72 to 1.1]

22. Secondary Outcome: Renal Clearance on Cycle 1 Day 21
Description: Renal clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by the kidneys.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle 1 Day 21
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 5 | 3 | 3 | 2 | 5 | 4
L/hour | 0.623 (NA) — Not reported when the number of participants is 2 or less. | 1.36 (42) | 0.754 (41) | 0.385 (42) | 1.14 (79) | 0.403 (53) | 1.27 (60) | 1.21 (NA) — Not reported when the number of participants is 2 or less. | 0.666 (27) | 1.08 (132)

23. Secondary Outcome: Amount of Unchanged Drug Excreted in Urine (Over the Dosing Interval) on Cycle 1 Day 21
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle 1 Day 21
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (mcg)
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 5 | 3 | 3 | 2 | 5 | 4
microgram (mcg) | 352 (NA) — Not reported when the number of participants is 2 or less. | 1027 (15) | 1933 (43) | 2357 (91) | 8524 (63) | 9066 (44) | 30180 (46) | 27710 (NA) — Not reported when the number of participants is 2 or less. | 44570 (38) | 77770 (85)

24. Secondary Outcome: Percentage of Dose Excreted Unchanged in Urine (Over the Dosing Interval) on Cycle 1 Day 21
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle 1 Day 21
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 5 | 3 | 3 | 2 | 5 | 4
Percentage of dose | 7.03 (NA) — Not reported when number of participants is 2 or less. | 10.3 (15) | 9.68 (43) | 5.89 (91) | 10.7 (63) | 7.57 (44) | 16.8 (46) | 10.3 (NA) — Not reported when number of participants is 2 or less. | 11.1 (38) | 13.0 (85)

25. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based on assessment of disease response according to disease specific response criteria (hematologic, cytogenetic and molecular responses). Results were analyzed based on malignancies, according to the planned analysis.
Time Frame: Baseline to end of study (up to 537 days)
Population: The Efficacy Analysis Set consisted of all enrolled participants who received Cycle 1 Day 1 dose of PF-04449913.
Measure: Number; unit: Percentage of participants
Groups:
- MDS and CMML: Participants with myelodysplastic syndrome (MDS)/chronic myelomonocytic leukemia (CMML) received oral single agent PF-04449913 tablets (5, 10, 20, 40, 80, 120, 180, 270, 400 or 600 mg) once on Day -6 (as a lead-in dose), followed by QD dosing starting on Cycle 1 Day 1, without interruption, in 28-day cycles.
- Myelofibrosis: Participants with myelofibrosis received oral single agent PF-04449913 tablets once (5, 10, 20, 40, 80, 120, 180, 270, 400 or 600 mg) on Day -6 (as a lead-in dose) followed by QD dosing starting on Cycle 1 Day 1, without interruption, in 28-day cycles.
- Acute Myeloid Leukemia: Participants with acute myeloid leukemia received oral single agent PF-04449913 tablets (5, 10, 20, 40, 80, 120, 180, 270, 400 or 600 mg) once on Day -6 (as a lead-in dose), followed by QD dosing starting on Cycle 1 Day 1, without interruption, in 28-day cycles.
- Chronic Myeloid Leukemia (Accelerated Phase/Blast Crisis): Participants with chronic myeloid leukemia (accelerated phase/blast crisis) received oral single agent PF-04449913 tablets (5, 10, 20, 40, 80, 120, 180, 270, 400 or 600 mg) once on Day -6 (as a lead-in dose), followed by QD dosing starting on Cycle 1 Day 1, without interruption, in 28-day cycles.
- Chronic Myeloid Leukemia (Chronic Phase): Participants with chronic myeloid leukemia (chronic phase) received oral single agent PF-04449913 tablets (5, 10, 20, 40, 80, 120, 180, 270, 400 or 600 mg) once on Day -6 (as a lead-in dose), followed by QD dosing starting on Cycle 1 Day 1, without interruption, in 28-day cycles.
Arm/Group | MDS and CMML | Myelofibrosis | Acute Myeloid Leukemia | Chronic Myeloid Leukemia (Accelerated Phase/Blast Crisis) | Chronic Myeloid Leukemia (Chronic Phase)
Number analyzed (Participants) | 7 | 7 | 28 | 2 | 2
Percentage of participants | 28.6 | 28.6 | 32.1 | 0 | 0

26. Secondary Outcome: Time to Progression (TTP)
Description: Time in months from start of study treatment to first documentation of objective disease progression or death due to cancer, whichever comes first. TTP was calculated as (first event date - date of first dose of study medication + 1)/30.4. Disease progression was determined from oncologic assessment data (where data met the criteria for disease progression: categorized as early progressor from chronic phase [CP], progressor to accelerated phase [AP] or blast crisis [BC] from CP or return to CP, progressor to AP to BC, loss of confirmed complete hematologic response, or loss of major cytogenetic response).
Time Frame: Baseline to end of study, up to 36 months
Population: The Efficacy Analysis Set consisted of all enrolled participants who received Cycle 1 Day 1 dose of PF-04449913.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MDS and CMML | Myelofibrosis | Acute Myeloid Leukemia | Chronic Myeloid Leukemia (Accelerated Phase/Blast Crisis) | Chronic Myeloid Leukemia (Chronic Phase)
Number analyzed (Participants) | 7 | 7 | 28 | 2 | 2
months | NA [1.84 to NA] — Median and upper limit of 95% confidence interval (CI) was not achieved/estimable due to the limited number of participants with events in the study. | 10.12 [2.79 to NA] — Upper limit of 95% CI was not achieved/estimable due to the limited number of participants with events in the study. | 2.83 [0.99 to 6.47] | 3.75 [NA to NA] — 95% CI was not achieved/estimable due to the limited number of participants with events in the study. | NA [NA to NA] — Median and 95% CI were not achieved/estimable due to the limited number of participants with events in the study.

27. Secondary Outcome: Duration of Response (DR)
Description: Time in months from the first documentation of objective response to objective disease progression or death due to any cancer. DR was calculated as [date of first documentation of progression or death due to cancer - date of first disease response + 1]/30.4. DR was calculated for the subgroup of participants with an objective disease response.
Time Frame: Baseline to end of study, up to 36 months
Population: The Efficacy Analysis Set consisted of all enrolled participants who received Cycle 1 Day 1 dose of PF-04449913.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Chronic Myeloid Leukemia (Chronic Phase): Participants with chronic phase chronic myeloid leukemia received oral single agent PF-04449913 tablets (5, 10, 20, 40, 80, 120, 180, 270, 400 or 600 mg) once on Day -6 (as a lead-in dose), followed by QD dosing starting on Cycle 1 Day 1, without interruption, in 28-day cycles.
Arm/Group | MDS and CMML | Myelofibrosis | Acute Myeloid Leukemia | Chronic Myeloid Leukemia (Accelerated Phase/Blast Crisis) | Chronic Myeloid Leukemia (Chronic Phase)
Number analyzed (Participants) | 7 | 7 | 28 | 2 | 2
months | 21.45 [NA to NA] — 95% CI was not achieved/estimable due to the limited number of participants with events in the study. | NA [3.71 to NA] — Median and upper limit of 95% CI were not achieved/estimable due to the limited number of participants with events in the study. | 2.83 [1.41 to 3.75] | NA [NA to NA] — Median and 95% CI were not achieved/estimable due to the limited number of participants with events in the study. | NA [NA to NA] — Median and 95% CI were not achieved/estimable due to the limited number of participants with events in the study.

28. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time in months from start of study treatment to first documentation of objective disease progression or death due to any cause. PFS was calculated as [first event date - date of first dose of study medication + 1]/30.4. Disease progression was determined from oncologic assessment data (where data met the criteria for disease progression: categorized as early progressor from CP, progressor to AP or BC from CP or return to CP, progressor to AP to BC, loss of confirmed complete hematologic response, or loss of major cytogenetic response; or from adverse event data (where the outcome was "Death").
Time Frame: Baseline to end of study, up to 36 months
Population: The Efficacy Analysis Set consisted of all enrolled participants who received Cycle 1 Day 1 dose of PF-04449913.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MDS and CMML | Myelofibrosis | Acute Myeloid Leukemia | Chronic Myeloid Leukemia (Accelerated Phase/Blast Crisis) | Chronic Myeloid Leukemia (Chronic Phase)
Number analyzed (Participants) | 7 | 7 | 28 | 2 | 2
months | NA [1.84 to NA] — Median and upper limit of 95% CI were not achieved/estimable due to the limited number of participants with events in the study. | 4.43 [2.07 to NA] — Upper limit of 95% CI was not achieved/estimable due to the limited number of participants with events in the study. | 2.83 [0.99 to 3.75] | 3.75 [NA to NA] — 95% CI was not achieved/estimable due to the limited number of participants with events in the study. | NA [NA to NA] — Median and 95% CI were not achieved/estimable due to the limited number of participants with events in the study.

29. Secondary Outcome: Number of Participants With Increase From Baseline in Corrected QT Interval Using Fridericia's Formula (QTcF)
Description: Triplicate 12-lead electrocardiogram (ECG) measurements (each recording separated by approximately 2 minutes) were performed and the average was calculated. The time from ECG Q wave to the end of the T wave corresponding to electrical systole (QT) was corrected for heart rate (QTc). QTc using Fridericia's formula (QTcF) was calculated. Participants with maximum increase from baseline of <30 millisecond (msec), 30 to <60 msec and >=60 msec were summarized.
Time Frame: Screening; predose, 1, 4, 24 hours (hr) postdose on Day -6; predose, 1 hr postdose on Cycle 1 Day 1; 1 hr postdose on Cycle 1 Days 8, 15; Day 1 of every subsequent cycle; predose, 1, 2, 4, 24 hr postdose for Cycle 1 Day 21; EOT (max reached: Cycle 20)
Population: QTc analysis set included all enrolled participants who had at least 1 ECG assessment after receiving at least 1 dose of PF-04449913.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5
Participants
  QTcF, maximum increase from baseline: <30 msec | 2 | 3 | 3 | 4 | 7 | 2 | 1 | 2 | 2 | 0
  QTcF, maximum increase from baseline: 30-<60 msec | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 3 | 7 | 0
  QTcF, maximum increase from baseline: >=60 msec | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5

30. Secondary Outcome: Number of Participants With Decrease From Baseline in QTcF Interval
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and the average was calculated. QTcF was calculated. Participants with maximum decrease from baseline of <30 msec, 30 to <60 msec and >=60 msec were summarized.
Time Frame: Baseline up to maximum of 537 days
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5
Participants
  QTcF, maximum decrease from baseline: <30 msec | 1 | 2 | 2 | 1 | 5 | 2 | 3 | 1 | 9 | 4
  QTcF, maximum decrease from baseline: 30-<60 msec | 1 | 1 | 2 | 3 | 3 | 0 | 0 | 2 | 0 | 0
  QTcF, maximum decrease from baseline: >=60 msec | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

31. Secondary Outcome: Number of Participants With Post-baseline QTcF Interval >= 500 Msec
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and the average was calculated. QTcF was calculated. Participants with post-baseline absolute QTcF values >=500 msec were summarized.
Time Frame: Baseline up to maximum of 537 days
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 8 | 3 | 3 | 5 | 9 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04449913 5 mg | PF-04449913 10 mg | PF-04449913 20 mg | PF-04449913 40 mg | PF-04449913 80 mg | PF-04449913 120 mg | PF-04449913 180 mg | PF-04449913 270 mg | PF-04449913 400 mg | PF-04449913 600 mg
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 2/4 | 3/4 | 5/8 | 2/3 | 2/3 | 3/5 | 8/9 | 3/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 4/4 | 8/8 | 3/3 | 3/3 | 5/5 | 9/9 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04449913 5 mg (N=3) | PF-04449913 10 mg (N=3) | PF-04449913 20 mg (N=4) | PF-04449913 40 mg (N=4) | PF-04449913 80 mg (N=8) | PF-04449913 120 mg (N=3) | PF-04449913 180 mg (N=3) | PF-04449913 270 mg (N=5) | PF-04449913 400 mg (N=9) | PF-04449913 600 mg (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 1
Pneumonal fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04449913 5 mg (N=3) | PF-04449913 10 mg (N=3) | PF-04449913 20 mg (N=4) | PF-04449913 40 mg (N=4) | PF-04449913 80 mg (N=8) | PF-04449913 120 mg (N=3) | PF-04449913 180 mg (N=3) | PF-04449913 270 mg (N=5) | PF-04449913 400 mg (N=9) | PF-04449913 600 mg (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 0 | 3 | 0 | 0 | 1 | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 5 | 0 | 0 | 1 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 3 | 2
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 2 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 3 | 4 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 3 | 1 | 5 | 2
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Tongue haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 1 | 3 | 1
Asthenia (General disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Condition aggravated (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Crepitations (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 2 | 1
Impaired healing (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 2 | 2 | 1 | 0 | 1 | 3 | 2
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 3 | 1 | 0
Spinal pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Albumin urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure diastolic decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Monocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 1 | 2 | 1 | 2 | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 4 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 1 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 2 | 3 | 0 | 1 | 1 | 3 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 5 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penile blister (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 1 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nail discomfort (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blue toe syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Some participants were administered the lead-in dose at other times (other than Day -6 as stated) due to changes in the timing of the lead-in dose as the protocol was amended a few times.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.